CLINICAL TRIAL: NCT02791893
Title: Vagus Nerve Stimulation: A Non-invasive Treatment to Improve the Health of Gulf Veterans With Gulf War Illness
Brief Title: Vagus Nerve Stimulation: Treatment for Gulf Veterans With Gulf War Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benjamin Natelson (Other)
Responsible Party: Sponsor-Investigator, Benjamin Natelson, Professor of Neurology, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 16-0350
Record Dates: First submitted 2016-05-30; First posted 2016-06-07 (Estimated); Results first posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Pain; Migraine
MeSH Terms: conditions — Pain; Migraine Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- VNS device (Experimental): Vagus Nerve Stimulation (VNS) hand held device - subjects to utilize the VNS hand held device for 20 weeks total, putting it on the skin overlying the vagus nerve in their neck and then turning it on for 120 second periods three times a day. The device is programmed to deliver only 6 bouts of stimulation per day - one to each side of the neck three times a day
  Interventions: Device: VNS device
- Inactive device (Placebo Comparator): Inactive hand held device - subjects to utilize the inactive device for 10 weeks and then will receive the VNS device for the next 10 weeks.
  Interventions: Device: VNS device; Device: Inactive device

INTERVENTIONS:
Device: VNS device — Hand held device to use for self administration of vagus nerve stimulation.
  Other Names: Non-InvasiveVagus Nerve Stimulation (nVNS) Therapy
Device: Inactive device — Hand held device to use for self administration of simulated vagus nerve stimulation.
  Arms: Inactive device

SUMMARY:
The researchers propose studying Gulf veterans with Gulf War Illness (GWI), characterized by a problem with widespread pain. Besides their pain, the researchers will also assess the effect of vagus nerve stimulation (VNS) in alleviating migraine headache, another complaint of Gulf veterans, which is common in the presence of widespread pain. Importantly, the researchers are partnering with a company that has made a hand-held device that allows for stimulation of the vagus nerve without the need for surgery; it works by the patient putting it on the skin overlying the vagus nerve in their neck and then turning it on for 120 second periods three times a day. The device is programmed to deliver only 6 bouts of stimulation per day - one to each side of the neck three times a day; it is then inactive until the next day. The fact that this device can be used without surgery and is non-invasive makes it extremely practical for use.

After collecting pre-treatment measurement of pain severity and headache severity, veterans will receive either the actual active VNS device or an inactive device, which does not stimulate the nerve. Veterans will use their device for ten weeks - providing similar information periodically over this period by responding to questions about the severity of their pain and headaches, They will then return to the Center for the final phase of the study where all veterans will receive active devices. Ten weeks later, they will return to the Center to provide information to allow the investigators to gain further knowledge as to the effectiveness of actual VNS in relieving pain - both throughout the body and in the head.

DETAILED DESCRIPTION:
The Three Phases of the Study

Subject Identification Phase of Study face to face visit at the War Related Illness & Injury Study Center at the East Orange Veterans Administration Medical Center (EOVAMC).

Blinded Phase of Study Office Visit [first time at Icahn School of Medicine at Mount Sinai. (ISMMS)] Subjects randomized to either VNS device or inactive device.

Open Label Phase of Study All subjects receive the VNS device

ELIGIBILITY:
Inclusion Criteria:

To be eligible for enrollment in the Study, patients must meet all of the following criteria:

* Patient is a veteran of the 1990-91 Gulf War, aged at least 42 years old
* Patient fulfills Kansas criteria for Gulf War Illness including endorsement of musculoskeletal pain at moderate or severe intensities. This means patient has endorsed symptoms in at least 3 of the following problem areas: Fatigue/sleep; musculoskeletal pain; cognitive and mood; Gastrointestinal; respiratory; skin.
* Patient has widespread pain as evidenced by endorsement of pain in at least 3 bodily quadrants plus in the axial skeleton
* Patient has a median 24 hour widespread pain score of at least 5 on a 0 to 10 visual analog scale (VAS) with data taken on five days
* To be considered as having migraine, the patient must fulfill International Headache Society (IHS) criteria, and it should have been present for at least one year prior to entry into the study
* Patient agrees to use the study device as intended, follow all of the requirements of the study including completion of diary after each self-treatment, follow-up visit requirements, complete self assessment questionnaires as scheduled, and report any adverse device effects to the study center within 24 hours of such adverse device effect.
* Patient is able to provide written Informed Consent.

Exclusion Criteria:

Patients with any of the following will not be eligible for enrollment:

* Patient has a history of intracranial aneurysm, intracranial hemorrhage, brain tumor or significant head trauma.
* Patient has in the opinion of the investigator a clinically relevant structural abnormality at the gammaCore-R treatment site (e.g., neoplasm, lymphadenopathy, previous surgery, neoplasm or abnormal anatomy).
* Patient has pain at the gammaCore treatment site (eg, dysesthesia, neuralgia, cervicalgia).
* Patient has other significant pain problem (e.g., cancer pain or other head or facial pain disorder) that in the opinion of the investigator may confound the study assessments.
* Patient has known or suspected severe cardiac disease (e.g., symptomatic coronary artery disease, prior myocardial infarction, congestive heart failure (CHF), significant premature ventricular contraction) or a history of cardiac arrhythmia.
* Patient has known or suspected cerebrovascular disease (e.g., prior stroke or transient ischemic attack, symptomatic carotid artery disease, prior carotid endarterectomy or other vascular neck surgery).
* Patient's electrocardiogram shows evidence of heart disease or arrhythmia including an abnormal baseline ECG (e.g. second and third degree heart block, prolonged QT interval (corrected QT (QTcB) interval >470 msec for women and > 450 for men), atrial fibrillation, atrial flutter, history of ventricular tachycardia or ventricular fibrillation, or clinically significant premature ventricular contraction) or a history of cardiac arrhythmia.
* Patient has had a previous cervical vagotomy.
* Patient has uncontrolled high blood pressure (systolic bp >160, or diastolic bp > 100) after 3 measurements within 24 hours.
* Patient is currently implanted with an electrical and/or neurostimulator device (e.g. cardiac pacemaker or defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant, Sphenopalatine ganglion stimulator or Occipital nerve stimulator).
* Patient has been implanted with metal cervical spine hardware or has a metallic implant near the gammaCore-R stimulation site.
* Patient has a history of significant syncope within the last 5 years.
* Patient has a history of non-epileptic or epileptic seizures within the last 5 years.
* Patient, in the opinion of the investigator, has a known history or suspicion of substance abuse or addiction within the last 5 years.
* Patient, in the opinion of the investigator/research staff, the patient is incapable of operating the gammaCore-R device as intended and performing the data collection procedures.
* Patient has a psychiatric or cognitive disorder and/or behavioral problem which in the opinion of the clinician may interfere with the study (e.g. Bipolar Disorder, depressive disorder with psychotic features, Specific Phobia, Acute Stress Disorder).
* Patient is pregnant or thinking of becoming pregnant in the next 6 months, or is of childbearing years and unwilling to use an accepted form of birth control or is unwilling to undergo pregnancy testing.
* Patient is nursing
* Patient has undergone botulinum toxin (BOTOX) injections of the head and/or neck in the last 3 months.
* Patient is participating or has participated in any other therapeutic clinical investigation during the last 30 days.
* Patient belongs to a vulnerable population or has any condition such that his or her ability to provide informed consent, comply with follow-up requirements, or provide self-assessments is compromised (e.g., homeless, developmentally disabled, prisoner).
* Patient has evidence of suicidality based on the Columbia Suicide Screening test
* Patient has previously used a gammaCore device.
* Patient is the spouse or housemate of someone else in the trial.

Ages: 42 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin H Natelson, MD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (4):
- United States (4):
  - East Orange Veterans Administration Medical Center, East Orange, New Jersey
  - Mount Sinai Beth Israel, New York, New York
  - Pain and Fatigue Study Center - Beth Israel Medical Center, New York, New York
  - Pain and Fatigue Study Center - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We started with 29 veterans, recruited at the East Orange VA, who agreed to participate. Of these, 27 actually came to the Icahn School of Medicine at Mount Sinai where they signed an informed consent and were randomized. From that sample, 20 veterans completed the blinded phase of the study and 15 completed the entire study including open trial.
Period: Blinded Phase
Arm/Group | VNS Device | Inactive Device
Started | 13 | 14
Completed | 10 | 10
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2
Period: Open Label Phase
Arm/Group | VNS Device | Inactive Device
Started | 10 | 10
Completed | 7 | 8
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VNS Device | Inactive Device | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.92 (7.11) | 55.46 (5.72) | 54.19 (6.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 12 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 9 | 12 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 7 | 10 | 17
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27
Pain Visual Analog Scale (0-10) [Mean (Standard Deviation); unit: units on a scale] — Patients used the Pain Visual Analog Scale (0-10; 0=No pain, 10=Worst pain possible) to rate their average level of pain over the last 24 hours. The median value for each individual's rating over 5 consecutive days immediately prior to the baseline was recorded and then the average was calculated for each group.
  units on a scale | 6.23 (0.73) | 6.82 (1.23) | 6.54 (1.05)
Physical Function Subscale from the Short Form Health Survey (SF-36) [Mean (Standard Deviation); unit: Normalized units on a scale] — A normalized indicator of physical functioning with a range from 0-100. Higher scores indicate fewer limitations to activity.
  Normalized units on a scale | 46.15 (22.28) | 40.00 (22.01) | 42.96 (21.94)
Number of Headache Days collected from the Migraine Disability assessment (MIDAS) [Mean (Standard Deviation); unit: Days] — Participants are asked to indicate the number of days in the last 3 months during which they experienced a headache. If a headache lasted more than 1 day, they are instructed to count each day. Scores are expected between 0-90 with higher numbers corresponding to a greater number of headache days.
  Days | 8.38 (9.59) | 14.21 (24.28) | 11.41 (18.60)
Depression subscale from the Hospital Anxiety and Depression Scale (HADS) [Mean (Standard Deviation); unit: Units on a scale] — A 14-item scale intended to quantify symptoms of depression and anxiety. Scores range from 0-21 on each subscale (Anxiety and Depression) with higher scores indicating a greater number of symptoms.
  Units on a scale | 9.46 (2.26) | 11.00 (1.88) | 10.26 (2.18)

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) to Assess Change of Widespread Pain
Description: Patients used the Pain Visual Analog Scale (0-10; 0=No pain, 10=Worst pain possible) to rate their average level of pain over the last 24 hours. The median value for each individual's ratings over 5 consecutive days immediately prior to the end of the intervention period was recorded and then the average was calculated for each group.
Time Frame: 10 and 20 weeks
Population: The 10-week measure includes only those individuals who completed the blinded phase of the study. The 20-week measure includes only those individuals who completed the open label phase of the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | VNS Device | Inactive Device
Number analyzed (Participants) | 10 | 10
Units on a scale
  10 weeks | 4.70 (2.41) | 5.40 (2.27)
  20 weeks: number analyzed (Participants) | 7 | 8
  20 weeks | 5.43 (2.07) | 3.56 (1.40)
Statistical Analysis 1: Comparison: VNS Device vs Inactive Device; A power analysis was conducted with G*Power, specifying a standard Type I error (α = .05) and desired power of .80. Results indicated that a total sample of 26 would be sufficient. Below are the results of the intent-to-treat analysis. Patients that did not complete the assessment after the blinded phase had their baseline scores carried forward. Post-intervention pain severity was regressed on pre-intervention pain severity and condition, using an ANCOVA model; Test type: Superiority; p = 0.47, ANCOVA — The a priori threshold for statistical significance was p = 0.05
Statistical Analysis 2: Comparison: VNS Device vs Inactive Device; Below are the results of the per protocol analysis. Patients that did not complete the assessment after the blinded phase are not included limiting the sample to 10 subjects in each condition (N=20). Post-intervention pain severity was regressed on pre-intervention pain severity and condition, using an ANCOVA model; Test type: Superiority; p = 0.58, ANCOVA — The a priori threshold for statistical significance was p = 0.05

2. Secondary Outcome: Patient Global Improvement of Change (PGIC)
Description: PGIC is a 7-point scale used to quantify a patient's rating of overall improvement. Patients rate their change from 1 (no change or gotten worse) to 7 (considerable improvement). Higher scores indicate greater improvement since starting the intervention.
Time Frame: 10 and 20 weeks
Population: The 10-week measure includes only those individuals who completed the blinded phase of the study. The 20-weel measure includes only those individuals who completed the open label phase of the study.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | VNS Device | Inactive Device
Number analyzed (Participants) | 10 | 10
Score on a scale
  10 weeks | 4.00 (2.06) | 3.11 (1.90)
  20 weeks: number analyzed (Participants) | 7 | 8
  20 weeks | 3.71 (1.98) | 5.37 (1.41)
Statistical Analysis 1: Comparison: VNS Device vs Inactive Device; A power analysis was conducted with G*Power, specifying a standard Type I error (α = .05) and desired power of .80. Results indicated that a total sample of 26 would be sufficient. Below are the results of the intent-to-treat analysis. Patients that did not complete the assessment after the blinded phase were assigned a score of "1" indicating no change in their condition. Post-intervention PGIC scores were compared between conditions; Test type: Superiority; p = 0.23, t-test, 2 sided — The a priori threshold for statistical significance was p = 0.05; This was an independent t-test comparing the conditions on their perception of change since starting the intervention
Statistical Analysis 2: Comparison: VNS Device vs Inactive Device; Below are the results of the per protocol analysis. Post-intervention PGIC scores were compared between conditions; Test type: Superiority; p = 0.23, t-test, 2 sided — The a priori threshold for statistical significance was p = 0.05; This was an independent t-test comparing the conditions on their perception of change since starting the intervention; Mean Difference (Final Values) = 1.1 — Condition difference = Active - Sham

3. Secondary Outcome: Physical Function Subscale From the Short Form Health Survey (SF-36)
Description: A normalized indicator of physical functioning with a range from 0-100. Higher scores indicate fewer limitations to activity.
Time Frame: 10 and 20 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | VNS Device | Inactive Device
Number analyzed (Participants) | 10 | 10
Score on a scale
  10 weeks | 65.50 (19.78) | 55.56 (24.81)
  20 weeks: number analyzed (Participants) | 7 | 8
  20 weeks | 60.71 (32.97) | 56.25 (27.35)
Statistical Analysis 1: Comparison: VNS Device vs Inactive Device; A power analysis was conducted with G*Power, specifying a standard Type I error (α = .05) and desired power of .80. Results indicated that a total sample of 26 would be sufficient. Below are the results of the intent-to-treat analysis. Patients that did not complete the assessment after the blinded phase had their baseline scores carried forward. Post-intervention physical function scores was regressed on pre-intervention physical function and condition, using an ANCOVA model; Test type: Superiority; p = 0.13, ANCOVA — The a priori threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = 12.88 — Condition difference = Active - Sham
Statistical Analysis 2: Comparison: VNS Device vs Inactive Device; Below are the results of the per protocol analysis. Patients that did not complete the assessment after the blinded phase had their baseline scores carried forward. Post-intervention physical function scores was regressed on pre-intervention physical function and condition, using an ANCOVA model; Test type: Superiority; p = 0.12, ANCOVA — The a priori threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = 10.5

4. Secondary Outcome: Number of Headache Days Collected From the Migraine Disability Assessment (MIDAS).
Description: Participants are asked to indicate the number of days in the last 3 months during which they experienced a headache. If a headache lasted more than 1 day, they are instructed to count each day. Scores are expected between 0-90 with higher numbers corresponding to a greater number of headache days.
Time Frame: 10 and 20 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | VNS Device | Inactive Device
Number analyzed (Participants) | 10 | 10
Days
  10 weeks | 4.10 (6.76) | 13.78 (23.49)
  20 weeks: number analyzed (Participants) | 7 | 8
  20 weeks | 6.29 (10.63) | 14.25 (25.58)
Statistical Analysis 1: Comparison: VNS Device vs Inactive Device; A power analysis was conducted with G*Power, specifying a standard Type I error (α = .05) and desired power of .80. Results indicated that a total sample of 26 would be sufficient. Below are the results of the intent-to-treat analysis. Patients that did not complete the assessment after the blinded phase had their baseline scores carried forward. Post-intervention headache days was regressed on pre-intervention headache days and condition, using an ANCOVA model; Test type: Superiority; p = 0.58, ANCOVA — The a priori threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -5.71 — Condition difference = Active - Sham
Statistical Analysis 2: Comparison: VNS Device vs Inactive Device; Below are the results of the per protocol analysis. Patients that did not complete the assessment after the blinded phase had their baseline scores carried forward. Post-intervention headache days was regressed on pre-intervention headache days and condition, using an ANCOVA model; Test type: Superiority; p = 0.49, ANCOVA — The a priori threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -9.8 — Condition difference = Active - Sham

5. Secondary Outcome: Depression Subscale From the Hospital Anxiety and Depression Scale (HADS)
Description: The HADS is a 14-item scale intended to quantify symptoms of depression and anxiety. Scores range from 0-21 on each subscale (Anxiety and Depression) with higher scores indicating a greater number of symptoms.
Time Frame: 10 and 20 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | VNS Device | Inactive Device
Number analyzed (Participants) | 10 | 10
Units on a scale
  10 weeks | 9.00 (2.26) | 10.11 (1.05)
  20 weeks: number analyzed (Participants) | 7 | 8
  20 weeks | 7.50 (1.05) | 9.75 (2.25)
Statistical Analysis 1: Comparison: VNS Device vs Inactive Device; A power analysis was conducted with G*Power, specifying a standard Type I error (α = .05) and desired power of .80. Results indicated that a total sample of 26 would be sufficient. Below are the results of the intent-to-treat analysis. Patients that did not complete the assessment after the blinded phase had their baseline scores carried forward. Post-intervention depression scores were regressed on pre-intervention depression scores and condition, using an ANCOVA model; Test type: Superiority; p = 0.18, ANCOVA — The a priori threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -1.42 — Condition difference = Active - Sham
Statistical Analysis 2: Comparison: VNS Device vs Inactive Device; Below are the results of the per protocol analysis. Patients that did not complete the assessment after the blinded phase had their baseline scores carried forward. Post-intervention depression scores were regressed on pre-intervention depression scores and condition, using an ANCOVA model; Test type: Superiority; p = 0.25, ANCOVA — The a priori threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -1.10 — Condition difference = Active - Sham

6. Primary Outcome: Visual Analog Scale (VAS) to Assess Change of Widespread Pain
Description: as for outcome 1
Time Frame: Baseline and 20 weeks
Population: Regardless of the original condition assignment, outcomes from baseline and after the open-label period are compared. All patients received at least 10 weeks of active VNS therapy.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | VNS Device
Number analyzed (Participants) | 20
Units on a scale
  Baseline | 6.18 (0.82)
  20 weeks: number analyzed (Participants) | 15
  20 weeks | 4.43 (1.94)
Statistical Analysis 1: Comparison: VNS Device; Regardless of original condition assignment, patients' 2.5-month pain scores at the end of the open label phase were compared to their baseline scores using a dependent samples t-test. Below are the results of the intent-to-treat analysis. Patients that did not complete the assessment after the open-label phase had their most recent score carried forward. All patients included in this comparison received at least 10 weeks of VNS therapy; Test type: Superiority; p = 0.004, t-test, 2 sided — The a priori threshold for statistical significance was p = 0.05; This was a dependent t-test comparing pre-intervention scores to the scores collected at the end of the open label phase
Statistical Analysis 2: Comparison: VNS Device; Regardless of original condition assignment, patients' 2.5-month pain scores at the end of the open label phase were compared to their baseline scores using a dependent samples t-test. Below are the results of the per protocol analysis. Patients that did not complete the assessment after the open-label phase were excluded. All patients included in this comparison received at least 10 weeks of VNS therapy; Test type: Superiority; p = 0.005, t-test, 2 sided — This was a dependent t-test comparing baseline scores to the scores collected at the end of the open label phase

ADVERSE EVENTS:
Time Frame: Patients were asked to provide reports on adverse events after the first week of the blinded phase (Week 1), at the end of the blinded phase (Week 11), and in the final week of the open label phase (Week 20). Adverse event monitoring for the sample took place over the course of 3 years (March, 2017 - March 2020).
Description: Adverse events were logged by description, date of occurrence, severity, and whether or not they were serious. Subjects were counted as having experienced a specific adverse event if they reported it at any of the three time points.
Arm/Group | VNS Device | Inactive Device
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/14
Other Adverse Events (participants affected / at risk) | 9/13 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VNS Device (N=13) | Inactive Device (N=14)
Chest pains occurred shortly after randomization (General disorders) | 1 (1) | 0 (0) — After randomization but before the first use of the VNS device, the patient started experiencing chest pains. Patient was admitted into the hospital overnight for testing. Results were negative. The event does not appear to be device related.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VNS Device (N=13) | Inactive Device (N=14)
Arrhythmia (Cardiac disorders) | 1 | 0
Burning/stinging sensation (General disorders) | 1 | 1
Dizziness (General disorders) | 0 | 1
Facial droops (Musculoskeletal and connective tissue disorders) | 1 | 1
Frequent stools (Gastrointestinal disorders) | 0 | 1
Headache (General disorders) | 1 | 3
Lightheadedness (General disorders) | 1 | 0
Lip droop/quiver (Musculoskeletal and connective tissue disorders) | 2 | 2
Metallic taste (General disorders) | 1 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscle tightness (General disorders) | 3 | 2
Numbness (General disorders) | 1 | 0
Pain/radiating pain (General disorders) | 1 | 2
Redness/irritation (Skin and subcutaneous tissue disorders) | 2 | 3
Small bumps (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling (General disorders) | 1 | 0
Tenderness (General disorders) | 2 | 1
Tingling sensation (General disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT02791893/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT02791893/ICF_001.pdf